CLINICAL TRIAL: NCT01689584
Title: Study of Family COsegregation of Nucleotide VARiants in the Panel of Genes to Validate Their Use in Genetic Counseling
Brief Title: COsegregation of VARiants in Panel of Genes
Acronym: COVAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2011-11
Record Dates: First submitted 2012-05-14; First posted 2012-09-21 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Gene Mutation-Related Cancer; Genetic Predisposition
Keywords: BRCA1; BRCA2; VUS; co-segregation; genetic counseling; PALB2; panel of genes
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Covar (Other)
  Interventions: Genetic: salivary kit

INTERVENTIONS:
Genetic: salivary kit — The saliva samples will be made of selected related (DNA).

SUMMARY:
The aim of the COVAR project is to classify reliably a maximum of VUS of the French database in order to use them for the genetic counseling. The results obtained through this study will have a major impact on clinical management of the patients and their families conducting in some cases to propose a prophylactic surgery.

DETAILED DESCRIPTION:
Originally, the COVAR study was designed to explore Variants of unknown biological significance (VUS) in BRCA1 (BReast Cancer 1) and BRCA2 (BReast Cancer 2) genes, which are the two major genes identified in hereditary breast and/or ovarian cancers. Since then the study has evolved, in parallel with the evolution of diagnosis, first introducing the PALB2 (Partner and localizer of BRCA2) gene explored in diagnosis since 2015 and now opening the study to all the genes of the panels performed in diagnosis in families with a genetic predisposition syndrome to cancers.

The French UMD (Universal Mutation Database)-BRCA1/2, accredited by the French National Cancer Institute, collects anonymous results of genetic tests performed by authorized French laboratories since 1995, giving a real-time vision of families carrying the same VUS. In september 2011, the French UMD-BRCA1/2 database comprised 706 different variants in 1,300 BRCA1 families and 1,089 different variants in 2,101 BRCA2 families. In April 2021, this database contained 1,651 different VSU for BRCA1, 3,015 different VUS for BRCA2, 471 different VUS for PALB2, 68 for RAD51C and 66 for RAD51D.

Since 2017, new genes have been explored in the diagnostic setting as they have been reported as predisposing factors for cancers. This list is constantly evolving (Moretta et al., 2018; Dhooge et al., 2020). Data collection for these genes is ongoing and a new database (FrOG) gathering all VUS and mutations identified in the French oncogenetic network has been set up. We have set up a consortium agreement at the end of 2020. This database gathers to date 12 genes and 11,912 different variants in more than 40,000 French families.

One of the key measurable parameters for classification of VUS as causal mutations is their co-segregation with the disease. The average size of French families is relatively small, the information of variant co-segregation limited to one family would not be significant. However, the compilation of co-segregation results obtained from several families will allow to obtain more precise and complete estimations of the probability of causality of a given variant.

The objective of the COVAR study (COsegregation VARiants) is to organize co-segregation studies of the VUS of the database UMD-BRCA1/2, in order to determine the causal or non-causal nature of these variants. To organize the variants by their clinical relevance, a grid with 5 classes has been used: 1=neutral, 2=likely neutral, 3=VUS, 4=likely causal, 5=causal. The VUS of classes 3 and 4 will be candidates to co-segregation studies because they cannot be used for the genetic counseling.

In the selected families the index case will invite the family members (affected and unaffected) to provide a sample of salivary fluid to test the presence of the VUS. The probability that a VUS is causal will be calculated from the cosegregation data using a Bayesian model. The results will be integrated in the multifactorial model described by D. Goldgar, model integrating different parameters as amino acid conservation, structural impact of the variant, co-occurrence with a pathogenic mutation, family history and tumor characteristics.

ELIGIBILITY:
Inclusion Criteria:

Index cases:

* A person carrying a gene variant class 3 or 4, present and selected in the families of national database of genetic group and cancer (GGC Unicancer) which identifies the variations of all genes from the panel of genes of all French laboratories.
* Age ≥ 18 years.
* Signed written inform consent "index case"

Related parties:

* Any relative of an index case with cancer
* Any relative without cancer related to an index case, retained by investigators, based on family structure and degree of related compared to the index case
* Age ≥ 18 years
* Information and signature of the informed consent "selected relatives"

Exclusion Criteria:

* Minors
* Persons deprived of liberty or under guardianship (including curators).
* Absence of signed written inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2012-07-02 (Actual); Primary Completion 2033-01-02 (Estimated); Study Completion 2034-01-02 (Estimated)

PRIMARY OUTCOMES:
Perform the co-segregation analysis of the selected VUS in the families in order to classify the maximum of variants in terms of their probability to be pathogenic | up to 15 years

SECONDARY OUTCOMES:
• Propose a standardized method to classify VUS that can be integrated into the already existing classification established in the UMD-BRCA1/2 database, with the main focus on variants of class 4 (probably causal) and class 3 (unknown significance). | up to 15 years
• Maximize the number of VUS (both pathogenic and neutral) having associated recommendations for clinical management of at-risk relatives that can be used to guide genetic counselling. | up to 15 years
Assess the penetrance of several class 3 and 4 VUS probably associated with moderate cancer risk, using collected phenotype/genotype data on extended pedigrees. | up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Dominique STOPPA-LYONNET, PU-PH, Study Chair — Institut Curie; Sandrine CAPUTO, PhD, Study Director — Institut Curie
Locations (57):
- France (54):
  - Institut Curie - Hopital Rene Huguenin, Saint-Cloud, Haut de Seine
  - CHU Amiens - Hôpital Nord, Amiens
  - ICO - Centre Paul Papin, Angers
  - Centre Hospitalier d'Angoulème, Angoulême
  - Institut Sainte-Catherine, Avignon
  - CHU Besançon, Besançon
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Jacques Coeur, Bourges
  - CHU Morvan de Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier Hôtel Dieu, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpital Civil de Colmar, Colmar
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Groupe Hospitalier La Rochelle-Ré-Aunis, La Rochelle
  - Hôpital Flaubert, Le Havre
  - Centre Oscar Lambret, Lille
  - Chru Lille, Lille
  - CHU Dupuytren, Limoges
  - Hospices Civils de Lyon, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU La Timone, Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Georges Renon, Niort
  - CHRU Caremeau, Nîmes
  - Hôpital de la Source, Orléans
  - Hôpital Saint-Antoine, Paris
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Hôpital Tenon, Paris
  - Hôpital Saint-Louis, Paris
  - HEGP, Paris
  - CHU La Milétrie, Poitiers
  - CHU de Reims, Reims
  - ICC Courlancy, Reims
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU de Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - ICO - Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Strasbourg Europe ICANS, Strasbourg
  - Hopital de Hautepierre - Hôpital Universitaire, Strasbourg
  - Institut Claudius Regaud - IUCT - Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - CH Simone VEIL, Troyes
  - Centre Hospitalier de Valence, Valence
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - CHU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
  - Institut Curie, Paris, Île-de-France Region
- CHU de Pointe à Pitre, Pointe-à-Pitre, Guadeloupe
- CHU de Fort de France, Fort-de-France, Martinique
- CHU Sud Réunion Saint-Pierre, Saint-Pierre, Reunion

REFERENCES:
- See also: French BRCA1 database — http://www.umd.be/BRCA1/
- See also: French BRCA2 database — http://www.umd.be/BRCA2/